CLINICAL TRIAL: NCT00286143
Title: Evaluation of Effects of Additional Fentanyl to Epidural Bupivacaine for Post-Thoracotomy Pain in Neonates on Perioperative Outcome
Brief Title: Effects of Additional Fentanyl to Epidural Bupivacaine for Post-Thoracotomy Pain in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Arjunan Ganesh, MBBS, Children's Anesthesiology Associates
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004-10-3988
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2009-09-16 (Estimated); Status verified 2009-09

CONDITIONS: Congenital Cystic Adenomatoid Malformation
MeSH Terms: conditions — Cystic Adenomatoid Malformation of Lung, Congenital | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): Fentanyl added to Bupivacaine via epidural catheter.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Fentanyl is added to epidural Bupivacaine to be administered to neonates having thoracotomy for lung resections.
  Other Names: Actiq®; Duragesic®; Fentora™; Ionsys™; Sublimaze®

SUMMARY:
The study exams whether adding an opioid to the epidural infusion of a local anesthetic in neonates will significantly improve the quality of the postoperative analgesia.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the best pain medication to be infused in the epidural catheter. At CHOP, the medication infused in the epidural catheter following a chest operation in neonates is a local anesthetic (bupivacaine). However, even with this continuous infusion, neonates still require multiple doses of intravenous opioids (i.e. morphine) because of persistent or constant pain. The administration of intravenous opioids in neonates can have many side effects, such as respiratory depression (reduced breathing rate), sedation, urinary retention (inability to pass urine), itching, nausea and vomiting It has been well documented that by adding a small dose of any opioid to a local anesthetic given through an epidural catheter, the feeling of postoperative pain can be significantly improved in older children and in adults. It is not known whether the addition of an opioid to a local anesthetic is beneficial in neonates. In this study, we are comparing the standard local anesthetic (bupivacaine) with a combination of bupivacaine and a small dose of an opioid (fentanyl).

This is a randomized study and the type of medication given into the epidural catheter will be chosen on the day of the operation by a random drawing (like flipping a coin). Your child could receive one of the following:

1. bupivacaine 0.1%
2. bupivacaine 0.1% with fentanyl 2mcg/ml Neither you nor your doctors will know which arm of the study your child is in. In case of emergency, the pharmacy can tell your doctor what medication your child is receiving.

ELIGIBILITY:
Inclusion Criteria:

1. Infants 0-6 months of age who require a thoracotomy for lung resection.
2. Parents accept the placement of an epidural catheter.

Exclusion Criteria:

1. Premature infants
2. Patients allergic to fentanyl and/or bupivacaine.
3. Known medical contraindications. -

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2005-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the difference in amount of Intravenous nalbuphine required after thoracotomy for lung resection in patients receiving epidural bupivacaine + fentanyl versus patients receiving epidural bupivacaine. | First 48 hours post-operatively

SECONDARY OUTCOMES:
1. Determine in two treatment groups the difference in pain scores as measured by the CRIES pain scale ,the length of stay,the incidence of side effects (respiratory depression, bradypnea, bradycardia and urinary retention). | 48 hours post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Arjunan Ganesh, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Ganesh A, Adzick NS, Foster T, Cucchiaro G. Efficacy of addition of fentanyl to epidural bupivacaine on postoperative analgesia after thoracotomy for lung resection in infants. Anesthesiology. 2008 Nov;109(5):890-4. doi: 10.1097/ALN.0b013e31818aa6cb. PMID 18946302